CLINICAL TRIAL: NCT04595630
Title: Diagnostic and Prognostic Value of Cardiac Biomarkers for Early Coronary Bypass Occlusion in Patients Undergoing Coronary Revascularization
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02257; ch20Berdajs
Record Dates: First submitted 2020-10-06; First posted 2020-10-20 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Coronary Bypass Graft Occlusion
Keywords: coronary artery bypass grafting (CABG); cardiac biomarkers; coronary revascularization; high-sensitivity cardiac troponin (hs-cTn); myocardial infarction (MI); Coronary Computed Tomography (CCT); early coronary bypass graft occlusion
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data collection from the hospital records — The clinical data from the patients enrolled in the study, such as the medical history, functional state, and EuroSCORE, and the hematological, basic renal, hepatic, and metabolic chemistry findings (including cTn as defined per the protocol), the operative data (operating time, blood loss, cardiopulmonary and cross-clamp time, number of arterial and venous grafts, the number of distal anastomoses, flow measured at all bypass grafts at the end of the intervention and the need for an assist device) and CCT scan data (at discharge from hospital facility) will be obtained from the hospital records. The data will be entered into a database.

SUMMARY:
This study is to evaluate the correlation between hs-cTn level as cardiac biomarker for ischemia and early graft occlusion as assessed by CCT in patients undergoing coronary bypass surgery.

DETAILED DESCRIPTION:
The early diagnosis of the periprocedural myocardial infarction (MI) due to the bypass graft occlusion is an important element, in order to introduce early therapeutic strategies. Invasive coronary angiography (CA) is the gold standard to evaluate the postoperative myocardial ischemia due to the graft occlusion. Since this procedure has several important risks, such as thromboembolic events, dissection, bleeding, and contrast dye-induced nephropathy, in daily clinical practice, only patients with strong clinical suspicion of early MI following coronary artery bypass grafting (CABG) undergo this invasive procedure. There is a clinical need for the development of safe and accurate non-invasive diagnostic approaches to assess the early coronary bypass graft occlusion and to predict the consequent MI. A new clinical approach for the identification of the early post-procedural graft occlusion in patients undergoing CABG surgery is the high-sensitivity cardiac troponin (hs-cTn) cut-off level. The peri-operative bypass occlusion will be assessed by a Coronary Computed Tomography (CCT) scan which is a widely available non-invasive approach that permits an accurate evaluation of coronary stenosis. This study is to evaluate the correlation between hs-cTn level as cardiac biomarker for ischemia and early graft occlusion as assessed by CCT in patients undergoing coronary bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients with isolated coronary bypass surgery

Exclusion Criteria:

* Patients withholding or lacking informed consent
* Patients requiring a concomitant procedure
* Exclusion criteria concerning the CCT scan
* Patients with known allergy to iodine-containing contrast agents
* Renal function impairment (serum creatinine >140 mmol/l; estimated glomerular filtration rate (GFR) <30 ml/min/1.73 m2).
* Pregnancy
* Unstable clinical state or severe heart failure
* Patients with registered MI and registered bypass occlusion in coronary angiogram
* Patients that didn't undergo a CCT prior to discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who will undergo isolated coronary bypass surgery at the University Hospital Basel.
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in hs-cTn level (ng/L) | Day 0 to discharge date (max 10 days)
  hs-cTn level following CABG to correlate between hs-cTn level as cardiac biomarker for ischemia and early graft occlusion as assessed by CCT

SECONDARY OUTCOMES:
All-cause mortality during hospital stay (death before discharge) | Day 0 to discharge date (max 10 days)
  All-cause mortality during hospital stay (death before discharge)
Cardiac-related mortality during hospital stay | Day 0 to discharge date (max 10 days)
  Cardiac-related mortality during hospital stay
Myocardial infarction during hospital stay | Day 0 to discharge date (max 10 days)
  Myocardial infarction during hospital stay
Surgical or percutaneous coronary re-intervention during hospital stay | Day 0 to discharge date (max 10 days)
  Surgical or percutaneous coronary re-intervention during hospital stay
Stroke rate during hospital stay | Day 0 to discharge date (max 10 days)
  Stroke rate during hospital stay
Incidence of major adverse cardiac and cerebrovascular events (MACCE) during hospital stay | Day 0 to discharge date (max 10 days)
  Incidence of major adverse cardiac and cerebrovascular events (MACCE) during hospital stay. MACCE is defined as a combined event of in-hospital mortality, stroke and myocardial infarction.

OTHER OUTCOMES:
All-cause mortality | During one-year and 36 months follow up
  All-cause mortality
Cardiac-related mortality | During one-year and 36 months follow up
  Cardiac-related mortality
Myocardial infarction | During one-year and 36 months follow up
  Myocardial infarction
Stroke | During one-year and 36 months follow up
  Stroke
Congestive heart failure requiring hospitalization | During one-year and 36 months follow up
  Congestive heart failure requiring hospitalization
Surgical or percutaneous coronary intervention | During one-year and 36 months follow up
  Surgical or percutaneous coronary intervention
Incidence of major adverse cardiac and cerebrovascular events (MACCE) | During one-year and 36 months follow up
  Incidence of major adverse cardiac and cerebrovascular events (MACCE)
Correlation between intraoperative flow measurements and incidence of early bypass occlusion | Day 0 to discharge date (max 10 days)
  Correlation between intraoperative flow measurements and incidence of early bypass occlusion
Changes in ECG (= changes in the ST segment), prone for myocardial ischemia, during in-hospital period | Day 0 to discharge date (max 10 days)
  Changes in ECG (= changes in the ST segment), prone for myocardial ischemia, during in-hospital period

CONTACTS AND LOCATIONS:
Overall Officials: Denis Berdajs, Prof. Dr. med., Principal Investigator — Department of Cardiac Surgery, University Hospital Basel
Locations (3):
- University Hospital Centre Zagreb, Zagreb, Croatia
- Wroclaw Medical University, Wroclaw, Borowska, Poland
- Department for Cardiac Surgery, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Salikhanov I, Koechlin L, Gahl B, Voehringer L, Reuthebuch O, Dimanski D, Mawad BM, Berdajs D. Survival, adverse events and management of silent in-hospital coronary bypass graft occlusion. Open Heart. 2025 Jul 7;12(2):e003368. doi: 10.1136/openhrt-2025-003368. PMID 40623893